CLINICAL TRIAL: NCT01149291
Title: A 18 Months, Post-marketing Observational Study to Follow-up Patients With End Stage Renal Disease Undergoing Hemodialysis, Receiving sVDRA's for Prevention and Treatment of Secondary Hyperparathyroidism
Brief Title: A Study to Follow-up Patients With End Stage Renal Disease Undergoing Hemodialysis, Receiving Selective Vitamin D Receptor Activator's for Prevention and Treatment of Secondary Hyperparathyroidism
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-314
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Secondary Hyperparathyroidism; End Stage Renal Disease
Keywords: high sensitivity C-reactive protein (hsCRP); cardiorenal; end stage renal disease (ESRD); Secondary hyperparathyroidism (SHPT); dialysis; paricalcitol; osteodystrophy; selective Vitamin D receptor activators (sVDRA); chronic kidney disease
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- End stage renal disease patients

SUMMARY:
The aim of this post-marketing observational study is to obtain further data on the long term use, safety and efficacy of selective Vitamin D Receptor Activator's as it is prescribed in the normal clinical setting and according to the approved Summary of Product Characteristics for the treatment of secondary hyperparathyroidism in hemodialysis patients in Turkey. The relation of the safety data to PTH (Parathyroid hormone) suppression over time will be evaluated. Also the number and incidence of hypercalcemia and hyperphosphatemia will be recorded.

DETAILED DESCRIPTION:
The scientific purpose of this study is to obtain data on the use of sVDRA(Selective Vitamin D Receptor Activator) in real-life clinical practice. This study will allow us to observe drug effectiveness in a distinct geography. Treatment effects, as well as maintenance of the results will be recorded for a 18 months period in order to obtain experience in the long term use of sVDRA(Selective Vitamin D Receptor Activator). Furthermore in the centers, additional blood parameter, hsCRP (high sensitivity C-reactive protein), will be examined as part of the clinical routine.

The primary aim of the study is:

* To assess percentage change in iPTH (intact parathyroid hormone) level monthly among hemodialysis patients with sHPT (secondary hyperparathyroidism) receiving sVDRA (Selective Vitamin D Receptor Activator) therapy.

Secondary aims are:

* To observe changes in commonly assessed biochemical parameters for bone and mineral metabolism (Ca (Calcium), P (Phosphorus), ALP (Alkaline phosphatase) and additionally hsCRP (high sensitivity C-reactive protein) as cardiovascular inflammatory marker.
* To evaluate routinely checked parameters like albumin, hemoglobin and dialysis adequacy (KT/V).
* To collect and evaluate data from all adverse events in order to establish the safety profile of sVDRA(Selective Vitamin D Receptor Activator) in daily clinical practice.
* To collect mortality data 6 months after 12 months of observational period or 6 months after drop out.

Patients will be followed for 12 months within the post-marketing observational study and will be checked for mortality data 6 months after this follow up period. The enrollment period should not exceed 6 months.

All demographic information will be summarized by using descriptive statistics and graphs. Laboratory levels will be assessed by using mean, median, minimum, maximum, standard deviation and percentages on visit basis. The mean differences on laboratory levels between visits will also be summarized by graphics and assessed by using percentages.

Alkaline phosphatase and hsCRP (high sensitivity C-reactive protein) levels will also be summarized by using descriptive statistics and graphs per visit.

sVDRA (Selective Vitamin D Receptor Activator) dose changes per visits will be summarized by descriptive statistics and graphs.

Mortality will be analyzed with life tables. By taking into account the primary and secondary aims of the study, to be able to achieve the therapeutic success on iPTH (intact parathyroid hormone) level changes with sVDRA (Selective Vitamin D Receptor Activator) treatment and perform mortality assessment in following 6 months and collect data regarding safety and efficacy of sVDRAs (Selective Vitamin D Receptor Activators) in long term use, it has been determined to enroll totally 510 patients from 30 sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients with secondary hyperparathyroidism in the presence of chronic kidney disease stage 5 and receiving hemodialysis who is treated with sVDRA's (Selective Vitamin D Receptor Activator) injection
* iPTH (intact parathyroid hormone) >300pg/ml, corrected serum Ca (Calcium) < 10.2 mg/dl, serum P (Phosphorus) < 6 mg/dl
* Male and female (not pregnant or not planning to be pregnant in the next 12 months) patients equal to or older than 18 years of age
* Signed Informed consent by subject
* Hypertensive and Diabetic subjects must be on an optimal and steady medication regimen for more than 30 days

Exclusion Criteria:

* Subject has known hypersensitivity and/or toxicity to vitamin D metabolites and/or other product ingredients
* Subject has participated in a clinical study within the last month
* If sVDRA's (Selective Vitamin D Receptor Activator) are contraindicated according to the SmPC (Summary of Product Characteristics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESRD (End Stage Renal Disease) patients undergoing hemodialysis who at the time of entry are receiving sVDRA's (Selective Vitamin D Receptor Activator) as it is prescribed in the normal clinical setting and according to the approved SmPC (Summary of Product Characteristics) for the prevention or treatment of secondary hyperparathyroidism.
Sampling Method: Non-Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To assess percentage change in iPTH (intact Parathyroid Hormone) level monthly among hemodialysis patients with SHPT (Secondary Hyperparathyroidism) receiving sVDRA (Selective Vitamin D Receptor Activator) therapy | 12 months

SECONDARY OUTCOMES:
Calcium, Phosphorus, ALP (Alkaline Phosphatase) | Month 0
Calcium, Phosphorus, ALP (Alkaline Phosphatase) | Month 1
Calcium, Phosphorus, ALP (Alkaline Phosphatase) | Month 2
Calcium, Phosphorus, ALP (Alkaline Phosphatase) | Month 3
Calcium, Phosphorus, ALP (Alkaline Phosphatase) | Month 4
Calcium, Phosphorus, ALP (Alkaline Phosphatase) | Month 5
Calcium, Phosphorus, ALP (Alkaline Phosphatase) | Month 6
Calcium, Phosphorus, ALP (Alkaline Phosphatase) | Month 7
Calcium, Phosphorus, ALP (Alkaline Phosphatase) | Month 8
Calcium, Phosphorus, ALP (Alkaline Phosphatase) | Month 9
Calcium, Phosphorus, ALP (Alkaline Phosphatase) | Month 10
Calcium, Phosphorus, ALP (Alkaline Phosphatase) | Month 11
Calcium, Phosphorus, ALP (Alkaline Phosphatase) | Month 12
Calcium, Phosphorus, ALP (Alkaline Phosphatase) | After early termination
Albumin, hemoglobin and dialysis adequacy (KT/V) | Month 0
Albumin, hemoglobin and dialysis adequacy (KT/V) | Month 1
Albumin, hemoglobin and dialysis adequacy (KT/V) | Month 2
Albumin, hemoglobin and dialysis adequacy (KT/V) | Month 3
Albumin, hemoglobin and dialysis adequacy (KT/V) | Month 4
Albumin, hemoglobin and dialysis adequacy (KT/V) | Month 5
Albumin, hemoglobin and dialysis adequacy (KT/V) | Month 6
Albumin, hemoglobin and dialysis adequacy (KT/V) | Month 7
Albumin, hemoglobin and dialysis adequacy (KT/V) | Month 8
Albumin, hemoglobin and dialysis adequacy (KT/V) | Month 9
Albumin, hemoglobin and dialysis adequacy (KT/V) | Month 10
Albumin, hemoglobin and dialysis adequacy (KT/V) | Month 11
Albumin, hemoglobin and dialysis adequacy (KT/V) | Month 12
Albumin, hemoglobin and dialysis adequacy (KT/V) | After early termination
hsCRP (High Sensitivity C-Reactive Protein) | Month 0
hsCRP (High Sensitivity C-Reactive Protein) | Month 3
hsCRP (High Sensitivity C-Reactive Protein) | Month 6
hsCRP (High Sensitivity C-Reactive Protein) | Month 9
hsCRP (High Sensitivity C-Reactive Protein) | Month 12
hsCRP (High Sensitivity C-Reactive Protein) | After early termination
Serious Adverse events | 18 months
Mortality data | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Gucuk, MD, Study Director — AbbVie
Locations (22):
- Turkey (Türkiye) (22):
  - Site Reference ID/Investigator# 37822, Antalya
  - Site Reference ID/Investigator# 68286, Antalya
  - Site Reference ID/Investigator# 40677, Antalya
  - Site Reference ID/Investigator# 85153, Istanbul
  - Site Reference ID/Investigator# 40672, Istanbul
  - Site Reference ID/Investigator# 40674, Istanbul
  - Site Reference ID/Investigator# 40678, Istanbul
  - Site Reference ID/Investigator# 40686, Istanbul
  - Site Reference ID/Investigator# 61585, Istanbul
  - Site Reference ID/Investigator# 63764, Istanbul
  - Site Reference ID/Investigator# 63765, Istanbul
  - Site Reference ID/Investigator# 63766, Istanbul
  - Site Reference ID/Investigator# 69973, Istanbul
  - Site Reference ID/Investigator# 63763, Izmir
  - Site Reference ID/Investigator# 48127, Izmir
  - Site Reference ID/Investigator# 64444, Karaman
  - Site Reference ID/Investigator# 40684, Kayseri
  - Site Reference ID/Investigator# 48132, Konya
  - Site Reference ID/Investigator# 68283, Kütahya
  - Site Reference ID/Investigator# 68281, Mersin
  - Site Reference ID/Investigator# 68282, Mersin
  - Site Reference ID/Investigator# 69974, Mersin

REFERENCES:
- See also: Related Info — http://rxabbvie.com